CLINICAL TRIAL: NCT01790607
Title: An Open-label, Single-dose,Intravenous Administration Study to Compare the Pharmacokinetics and Safety of ONO-2745/CNS 7056 in Subjects With Chronic Hepatic Impairment With Matching Healthy Subjects
Brief Title: An Open-label, Single-dose, Intravenous Administration Study of ONO-2745/CNS 7056 in Subjects With Chronic Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-2745IVU007
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Hepatic Impairment; Healthy
Keywords: Adult healthy subjects will be matched with individual subjects by age (± 5 years, gender, and BMI (± 15%)
MeSH Terms: conditions — Coitus | interventions — remimazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Subjects with moderate chronic hepatic impairment (Experimental): Single IV bolus of ONO-2745/CNS 7056 over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: ONO-2745 /CNS 7056
- Healthy subjects matched to moderate hepatic impaired subjects (Experimental): Single IV bolus of ONO-2745/CNS 7056 over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: ONO-2745 /CNS 7056
- Subjects with mild chronic hepatic impairment (Experimental): Single IV bolus of ONO-2745/CNS 7056 over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: ONO-2745 /CNS 7056
- Healthy subjects matched to mild hepatic impaired subjects (Experimental): Single IV bolus of NO-2745/CNS 7056 over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: ONO-2745 /CNS 7056
- Subjects with severe chronic hepatic impairment (Experimental): Single IV bolus of ONO-2745/CNS 7056 over 1 minute at 0.1 mg/kg body weight
  Interventions: Drug: ONO-2745 /CNS 7056

INTERVENTIONS:
Drug: ONO-2745 /CNS 7056

SUMMARY:
To evaluate and compare the pharmacokinetics and safety of ONO-2745/CNS 7056 in subjects with the hepatic impairment and matched healthy subjects.

DETAILED DESCRIPTION:
In Part One, 8 subjects with moderate hepatic impairment (Child Pugh Scale B) and 8 matched healthy subjects will be enrolled. In Part 2, 8 subjects with mild hepatic impairment (Child-Pugh Scale A) and 8 matched healthy subjects will be enrolled. In Part 3, 3 subjects with severe hepatic impairment (Child-Pugh Scale C) will be enrolled. Parts 2 and 3 will only be initiated if the criteria per protocol is met in Part One. The pharmacokinetics and safety profiles will be compared between hepatic impaired subjects and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years of age
* Negative test for the selected drugs of abuse at screening

Hepatic impaired subjects:

* Stable hepatic function and medication regimen for at least 28 days prior to check-in
* Degree of hepatic impairment will be determined by the Child-Pugh Scale

Exclusion Criteria:

* Clinical manifestation of any disease (except hepatic impaired subjects)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, including food, or other substance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To study the effect of hepatic impairment on the pharmacokinetics of ONO-2745/CNS 7045 by assessment of drug concentration through blood sample analysis | PK: Pre-dose to 4 hours post-dose
To study the effect of ONO-2745/CNS 7045 on the subjects with hepatic impairment by evaluating the safety parameters per protocol including labs, vitals and adverse events | Overall safety: Pre-dose to 7 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (3):
- United States (3):
  - Anaheim Clinical Site, Anaheim, California
  - Orlando Clinical Site, Orlando, Florida
  - South Miami Clinical Site, South Miami, Florida

REFERENCES:
- [Derived] Stohr T, Colin PJ, Ossig J, Pesic M, Borkett K, Winkle P, Struys MMRF, Schippers F. Pharmacokinetic properties of remimazolam in subjects with hepatic or renal impairment. Br J Anaesth. 2021 Sep;127(3):415-423. doi: 10.1016/j.bja.2021.05.027. Epub 2021 Jul 8. PMID 34246461